CLINICAL TRIAL: NCT07025525
Title: Clinical and Radiographic Evaluation of Ultrasonic Activated Irrigation Versus Non Activated Irrigation in Pulpectomy of Necrotic Primary Molars : A Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Naira Essam Farouk, Internal resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: dentistry Cairo university
Record Dates: First submitted 2025-06-07; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Pulpectomy Agents
Keywords: Primary molars; Irrigation activation within the canal
MeSH Terms: interventions — Sodium Hypochlorite; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention group 1 (Experimental): Ultrasonic activated sodium hypochlorite
  Interventions: Device: Ultrasonic activated sodium hypochlorite
- Intervention group 2 (Experimental): Ultrasonic activated saline
  Interventions: Other: Ultrasonic acivated saline
- Intervention group 3 (Experimental): Sodium hypochlorite
  Interventions: Other: Sodium Hypochlorite Solution
- Control group 4 (Active Comparator): Saline
  Interventions: Other: Saline

INTERVENTIONS:
Device: Ultrasonic activated sodium hypochlorite — Using ultrasonic-activated sodium hypochlorite in the canals of primary molars can significantly enhance root canal disinfection by improving the irrigant's penetration and effectiveness. Primary molars often have complex and irregular canal anatomies, which can limit the reach of traditional irrigation methods. Ultrasonic activation creates acoustic streaming and cavitation effects, allowing sodium hypochlorite to better dissolve organic tissue and disrupt bacterial biofilms, especially in hard-to-reach areas. This leads to more thorough cleaning, reduced microbial load, and potentially better clinical outcomes in pediatric endodontics
  Arms: Intervention group 1
Other: Ultrasonic acivated saline — using ultrasonic-activated saline within the canals of primary teeth lies in its ability to enhance mechanical debridement and improve irrigation effectiveness without the risks associated with stronger chemical agents. Although saline lacks inherent antimicrobial properties, ultrasonic activation generates acoustic streaming and cavitation, which help dislodge debris, disrupt biofilms, and clean intricate canal anatomy more efficiently than passive irrigation. This makes it a safer alternative in pediatric patients, minimizing the risk of cytotoxic effects or damage to developing permanent tooth buds while still improving cleaning outcomes.
  Arms: Intervention group 2
Other: Sodium Hypochlorite Solution — using sodium hypochlorite (NaOCl) within the canals of primary molars is its excellent antimicrobial and tissue-dissolving properties, which are essential for effective root canal disinfection. Primary molars often have complex and irregular canal systems that harbor bacteria and necrotic tissue. Sodium hypochlorite not only helps eliminate a broad spectrum of microorganisms but also dissolves organic debris, improving canal cleanliness and reducing the risk of post-treatment infection. When used in appropriate concentrations, it can significantly enhance the success of pulpectomy procedures in pediatric patients while maintaining safety.
  Arms: Intervention group 3
Other: Saline — Saline is commonly used as an irrigant in the root canal treatment of primary molars due to its excellent biocompatibility and safety profile. It is a non-toxic, isotonic solution that poses no risk to the surrounding periapical tissues, which is particularly important in primary teeth where root resorption and open apices are common. This minimizes the chance of damaging the underlying permanent tooth germ, a critical consideration in pediatric dentistry. Saline is also safe if accidentally extruded beyond the apex or ingested, making it a suitable choice for young children.
  Arms: Control group 4

SUMMARY:
This is a Clinical and Radiographic Evaluation of Canal Irrigation Using Ultrasonically Activated vs. Non-Activated Irrigants in Pulpectomy of Necrotic Primary Molars: A Randomized Clinical Trial" This study aims to compare the effectiveness of using ultrasonically activated irrigant versus non-activated irrigant in terms of clinical and radiographic success rates in the pulpectomy of necrotic primary molars, through a randomized clinical trial.

DETAILED DESCRIPTION:
Primary teeth are considered of great importance to children allowing their normal, healthy development and growth while preserving function, eating, speech and normal development of occlusion while preserving the space for permanent dentition and guide their eruption.

Pulpectomy of primary molar teeth is considered as reasonable treatment approach to ensure either normal shedding or long term survival of 1ry teeth as fully functional component in dental arch.

Treatment of necrotic primary teeth is complex due to anatomical and physiological characteristics and high no. of bacterial species present in endodontic infection.

Treatment success depend on the elimination of root canal infection which can be done mechanically and chemically to ensure the complete removal of bacterial canal infection.

Irrigation is a key part of successful root canal treatment. It has several important functions, the most important one that it has a washing effect and an antimicrobial/antibiofilm effect. Irrigation is also the only way to impact those areas of the root canal wall not touched by mechanical instrumentation.

Ultrasonic activation cause irrigant streaming and cavitation phenomena resulting in significantly improved debridement of canal spaces, disruption of biofilm and improved penetration of irrigant into dentinal tubules and reduces bacterial level improving prognosis and ability to seal.

This study has been conducted by only few researchers, and there is limited evidence supporting the effect of ultrasonic activation on irrigation.

So this study is conducted to compare the effect of ultrasonic activation of irrigation on success of pulpectomy versus that of non-activated irrigation

ELIGIBILITY:
Inclusion Criteria:

-

Clinical Criteria:

1. Children aged between 4 to 7 years' old
2. Children with deep caries involving pulp in primary molars
3. History of abscess, swelling or pus
4. Pain on percussion
5. Mobility grade 1

Radiographic criteria:

1. Root resorption due to abscess less that ⅔ of root
2. Periapical RL or furcation RL
3. Widening in PDL space or loss of lamina dura continuity

Exclusion Criteria:

* Clinical criteria: -

  1. Refusal of participation.
  2. Patient unable to attend to follow up
  3. Non-restorable tooth.
  4. Medically compromised patient.
  5. Uncooperative patient

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | 6 months
  Post operative pain assessments will be clinically , binary yes or no oral from patients word
Soft tissue pathology | 6 months
  This outcome will be measured clinically , binary yes or no by visual inspection
Pain on percussion | 6 months
  Will measured clinically , binary yes or no using back of mirror for percussion assessment
Pathological mobility | 6 months
  Will be assessed clinically , binary by yes or no using back of mirror and finger of one hand to check mobility

SECONDARY OUTCOMES:
Furcation or periapical pathology | 6 months
  Will be measured clinically by periapical radiograph binary yes or no the presence of Radiolucency
External or internal root resorption | 6 months
  Will be assessed by radiograph binary yes or no checking radiolucency

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry cairo university, Cairo, Egypt

REFERENCES:
- [Background] Singh R, Barua P, Kumar M, Safaya R, Monajemi H, Monajemi H. Effect of Ultrasonic Instrumentation in Treatment of Primary Molars. J Contemp Dent Pract. 2017 Sep 1;18(9):750-753. doi: 10.5005/jp-journals-10024-2120. PMID 28874635
- [Background] Virdee SS, Seymour DW, Farnell D, Bhamra G, Bhakta S. Efficacy of irrigant activation techniques in removing intracanal smear layer and debris from mature permanent teeth: a systematic review and meta-analysis. Int Endod J. 2018 Jun;51(6):605-621. doi: 10.1111/iej.12877. Epub 2017 Dec 22. PMID 29178166
- [Background] Kumar RS, Ankola AV, Sankeshwari RM, Hebbal M, Hampiholi V, Kumar S L, Deshpande AP, Choudhury AR, Pai Khot AJ. Effectiveness of various irrigant activation techniques on the penetration of sodium hypochlorite into lateral canals of mature permanent teeth: A systematic review and meta-analysis. Saudi Dent J. 2023 Jan;35(1):1-23. doi: 10.1016/j.sdentj.2022.12.004. Epub 2022 Dec 16. PMID 36817024
- [Background] Ahmed, H.M.A., 2014. Pulpectomy procedures in primary molar teeth. European Journal of General Dentistry, 3(01), pp.3-10
- [Background] Fabris AS, Nakano V, Avila-Campos MJ. Bacteriological analysis of necrotic pulp and fistulae in primary teeth. J Appl Oral Sci. 2014 Apr;22(2):118-24. doi: 10.1590/1678-775720130358. PMID 24676582